CLINICAL TRIAL: NCT06084065
Title: Feasibility and Effectiveness of a Ring-type Blood Pressure Measurement Device Compared With 24-hour Ambulatory Blood Pressure Monitoring Device: Pilot Study
Brief Title: Feasibility and Effectiveness of a Ring-type Blood Pressure Measurement Device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hae-young Lee, Head of Cardiology, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2305-064-1431
Record Dates: First submitted 2023-10-05; First posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Hypertension; Blood Pressure; Systolic Hypertension; Diastolic Hypertension; Essential Hypertension; Obstructive Sleep Apnea; Prehypertension
MeSH Terms: conditions — Hypertension; Isolated Systolic Hypertension; Essential Hypertension; Sleep Apnea, Obstructive; Prehypertension

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ring arm (Experimental)
  Interventions: Device: CART-I Plus

INTERVENTIONS:
Device: CART-I Plus — Photoplethysmography based ring-type blood pressure measurement device

SUMMARY:
The goal of this clinical trial is to evaluate the feasibility and effectiveness of a ring-type blood pressure measurement device compared to a 24-hour ambulatory blood pressure monitoring device in patients with hypertension or suspected hypertension. The main question it aims to answer is whether the 24-hour blood pressure measurement accuracy of the ring-type blood pressure monitor is similar to that of the 24-hour ambulatory blood pressure monitor. To participate, subjects must wear a ring blood pressure monitor and an ambulatory blood pressure monitor simultaneously for 24 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for 24-hour ambulatory blood pressure monitoring for diagnostic purposes among those suspected of having hypertension
2. Confirmed hypertensive patients scheduled for 24-hour ambulatory blood pressure monitoring for treatment purposes

   * Either criterion 1 or 2 are planned to be selected as study participants.

Exclusion Criteria:

* Participants who do not consent to the study
* Individuals with a Body Mass Index of 30 or above (there's a concern of measurement errors as the standard 24-hour ambulatory blood pressure cuffs may not fit well)
* Pregnancy
* Baseline heart disease patients: individuals with a history of hospitalization due to heart failure, valvular disease, or myocardial infarction
* Patients diagnosed with atrial fibrillation on a 12 lead EKG within the past 6 months
* End-stage renal disease (patients undergoing dialysis)
* Users of mobile phones that are not compatible with the test device (CART-I plus) used in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-07-13 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The average agreement between blood pressure measured with a 24-hour ambulatory BP measurement device and blood pressure measured with a ring-type BP measurement device during a subject's activity time. | Compare the blood pressure measured over 24 hours using a ring-type blood pressure monitor and 24-hour ambulatory blood pressure monitoring.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National Univesity Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Lee H, Park S, Kwon H, Cho B, Park JH, Lee HY. Feasibility and Effectiveness of a Ring-Type Blood Pressure Measurement Device Compared With 24-Hour Ambulatory Blood Pressure Monitoring Device. Korean Circ J. 2024 Feb;54(2):93-104. doi: 10.4070/kcj.2023.0303. Epub 2023 Dec 26. PMID 38196118